CLINICAL TRIAL: NCT04692519
Title: Duet 2.0: Starting the Conversation: A New Intervention Model to Stimulate Language Growth in Underserved Populations
Brief Title: Duet 2.0 Starting the Conversation: A New Intervention Model to Stimulate Language Growth in Underserved Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: William Penn Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 26412
Record Dates: First submitted 2020-12-16; First posted 2020-12-31 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Language Development; Language, Child; Early Intervention
Keywords: Language development; Low-income; Linguistically diverse; Culturally diverse
MeSH Terms: conditions — Language

STUDY DESIGN:
Intervention Model Description: Participants who are selected to participate in the intervention will be given access to videos containing the Duet intervention modules. We will ask families to watch one Duet module a week, if possible. They will have up to 3 months to complete the 6 modules. Intervention participants will be scheduled for follow-up data collection at 3 months, 6 months, and pending funding, 1-year after baseline.
  Participants who are in the delayed access control group will not have to complete the modules and will be scheduled for a 3-month, 6-month, and pending funding, a 1-year follow-up calls. They will have delayed access to the modules, which means that they will receive access to the module videos at their 6-month study session and will be offered the opportunity to contact the research team with any questions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator and postdoctoral fellow on the project will both be blind. Only the coordinator will know who is the in intervention group and who is in the delayed access group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Duet 2.0 intervention is comprised of six training modules, which include behavioral strategies, real-life and animated examples of high-quality early language interactions, and interactive scenarios. Modules were translated into Spanish. Participants will watch one Duet intervention module a week and have up to 3 months to complete all 6 modules. As intervention families review the modules on their own time at home, they will receive remote coaching from an assigned interventionist and weekly module-specific fidelity/comprehension questions. Interventionists will check-in weekly via phone or video (~30-60 minutes), whichever is more convenient for the family. During the check-in, interventionists will do teach-back about the module, guide the family on how to incorporate the strategies into their daily lives, and provide feedback. Intervention participants will be scheduled for follow-up data collection at 3 months, 6 months, and pending funding, 1-year after baseline.
  Interventions: Behavioral: Duet Language Intervention Modules
- Delayed Access (No Intervention): Participants who are in the delayed access control group will not have to complete the modules and will be scheduled for a 3-month, 6-month, and pending funding, a 1-year follow-up calls. They will have delayed access to the modules, which means that they will receive access to the module videos at their 6-month study session and will be offered the opportunity to contact the research team with any questions.

INTERVENTIONS:
Behavioral: Duet Language Intervention Modules — The Duet 2.0 intervention modules promote the following guiding principles that help build effective communication. Below are the 5 principles covered in the six Duet modules: 1) General Awareness: Awareness and knowledge of child development 2) Creating Opportunities: Opportunities for communication during everyday activities 3) Conversational Duets: Rhythmic and reciprocal early language interactions 4) Scaffolding: Providing just enough help to support child independence 5) Harmonizing: Using the strategies together. These modules, which include behavioral strategies, real-life and animated examples of high-quality early language interactions, and interactive scenarios. The modules were informed and narrated by community members and carefully designed to address specific needs of high-risk communities. The modules have also been translated into Spanish, making sure to encompass specific cultural and dialect needs. Translation accuracy was verified by a qualified Spanish translator.
  Arms: Intervention

SUMMARY:
Caregiver-child language interactions in the first three years of life predict early language development, school readiness, and academic achievement. Despite the importance of these factors, there are disparities in the frequency and quality of children's early language interactions. Although there is within-group variability, children from low-income families, on average, have fewer and lower-quality language experiences than their middle- or high-income peers. The current study addresses a need in the community for an early language intervention accessible to low-income families who speak Spanish. This study will build upon research conducted in a previous study, "Enhancing the Communication Foundation-The Duet Project", by piloting the English and Spanish modules with families through a light-touch, remote intervention delivery model. Temple University Health System's Department of Pediatrics will aid in identifying participants. Baseline and follow-up measures will be used to evaluate caregiver knowledge of child development, psychosocial perceptions, demographics, caregiver-child language interaction quality, and child language skills. It is hypothesized that dyads who receive the intervention will make greater gains in early interaction quality, knowledge of child development, and child language skills than the delayed-access control group. This work has the potential to shape early intervention design and implementation for people in underserved communities across the country.

DETAILED DESCRIPTION:
Objectives and Background

The purpose of this study is to determine whether Duet 2.0- a light-touch, public health model of remote intervention delivery 1) increases caregiver knowledge about children's language development, 2) improves caregiver-child language interaction quantity and quality, and 3) enhances children's language skills. It is hypothesized that dyads who receive the Duet 2.0 intervention will make greater gains in knowledge of child development, early interaction quality, and child language skills than the delayed-access control group. Secondary analyses will be conducted to examine if and how parent (e.g., self-efficacy) and child (e.g., child language abilities) characteristics relate to each other, baseline measures, and treatment outcomes.

Early language skills are fundamental to language, cognitive, and socioemotional development and are the single best predictors of later academic success. Caregiver-child language interactions in the first three years of life not only predict early language development, but also influence school readiness skills and academic achievement. High-quality early language interactions are characterized by rich and diverse vocabulary, responsive talk (i.e., language following the child's attention), decontextualized language (e.g., language beyond the here and now context, "Remember we went to a party last night"), communication foundation (e.g., use of verbal and gestural symbols, engaging in back-and-forth conversations), and question use. In fact, early reading outcomes are particularly contingent on strong language skills that go beyond and accompany strong decoding skills.

Despite the importance of these factors, there are large disparities in the frequency and quality of children's early language interactions. Although there is great within-group variability, children from low-income families on average have fewer and lower-quality language experiences than their middle- or high-income peers. Early disparities in language experiences can lead to gaps in language skills and academic achievement that persist into adulthood.

Duet 2.0 will adopt an innovative and scalable approach-remote delivery and coaching. This design reflects arguably the strongest evidence for successful intervention. Remote coaching and telehealth are becoming accepted models for public health intervention in domains like nutrition, fitness, heart health, and diabetes. There is also growing support for remote delivery parent and teacher training programs. For instance, remote coaching has effectively improved Head Start teachers' language and literacy practices. This intervention model has also been used successfully to promote mental health in parents of infants, train parents in domains such as child socioemotional development, and support language and communication in young children with autism.

With the support of the William Penn Foundation and the Bezos Family Foundation, the PIs spent three years designing and piloting a caregiver- implemented early language intervention program-The Duet Project: Early Engagement, Future Success. Using community-based participatory research (CBPR) framework with partners at the Maternity Care Coalition (MCC), the PIs created Duet training materials that are evidence-based and culturally sensitive.

Pilot work with Duet yielded promising findings despite low sample sizes. These preliminary results support the efficacy of the Duet modules. Duet participants included some Spanish speakers; however, all participants had to be able to receive services in English. This significantly limited recruitment-nearly 25% of infants and toddlers in Philadelphia are of Latino/Hispanic origin. Furthermore, the percent of Hispanic/Latino people living in poverty is disproportionately high-they make up 21% of the population living in poverty but only 14.4% of the total population.

Translating the Duet modules into Spanish and developing a more efficient delivery system will maximize their scalability and positive impact on low-SES families. Establishing an efficient communication foundation, will enhance language learning and literacy development with the goal of narrowing the achievement gap in future generations. Given the undeniably powerful link between early language competencies and later literacy skills, this intervention has the potential to have long-lasting and widespread benefits both at local and national levels.

Duet 2.0 Intervention and Data Collection

Prospective research participants will be identified and recruited through the Department of Pediatrics at Temple University Health System(TUHS) and possibly by sharing recruitment materials with local community organizations (e.g., Early Head Start centers). Participants will be recruited and screened. If they meet study requirements during screening, they will then be consented and enrolled. Families who are randomly selected into the intervention group will complete the modules at home on their own time and receive remote coaching from an interventionist or coach (terms used interchangeably). Families in the delayed-access control group will receive access to the modules at the end of the study, but will still complete data-collection sessions. Approximately once a week after enrollment, Interventionists will support the intervention-group families remotely in comprehending and implementing what they have learned from the modules. Interventionists may also be involved in remote data collection. All participants will be scheduled for follow-up data collection sessions via phone or video conference.

ELIGIBILITY:
Inclusion Criteria

* To be included in this study, Caregivers (Control and Intervention Groups)

Caregivers must:

1. Live in a zip code that is within a 30-mile radius of Weiss Hall at Temple University
2. Be 18;0 years of age or older
3. Be a parent or legal guardian of participating child
4. Speak English and/or Spanish (at least 80% of the time)
5. Read English and/or Spanish "well" or "very well"
6. Have weekly access to phone or internet
7. Have adequate visual abilities to participate in the study (per participant report)
8. Have no hearing impairment or loss (per participant report) OR if some hearing impairment or loss, have received amplification (e.g., hearing aid, cochlear implants) and speak spoken (e.g., not signed) language as their primary mode of communication (per participant report).
9. Qualify as Low-Socioeconomic Status (Low-SES), which is defined as, being at or below 200% of the Federal Poverty Guideline (FPG) and having no more than a 4-year college degree

   * To be included in this study, children (Control and Intervention Groups) must:

a. Be between 12 and 30 months at baseline b. Be Spanish and/or English learners (at least 80% of the time), as defined by c. Have already acquired verbal or non-verbal intentional language (e.g., gesture to get someone's attention and/or point to request and obtain a toy) and speak no more than three-word utterances (per caregiver report) d. Have adequate visual abilities to participate in the study (per caregiver report) e. Have no hearing impairment or loss (per caregiver report) OR if some hearing impairment or loss, have received amplification (e.g., hearing aid, cochlear implants) and be learning spoken (e.g., not signed) language as their primary mode of communication (per caregiver report).

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Caregiver-Child Language Interaction | Baseline, 3-month follow-up, and 6-month follow-up
  To assess the quality of caregiver-child interactions, caregivers and participating children will be filmed or film themselves for a total of 10-15 minutes, at baseline, 3-month, and 6-month follow-up sessions. We will calculate the number of conversational turns.
Change in Parent/Provider Expectations and Knowledge | Baseline, 3-month follow-up, and 6-month follow-up
  Caregiver's knowledge of child development will be assessed at baseline and post intervention. The Parent/Provider Expectations and Knowledge-II (SPEAK-II) is a well-validated measure used in similar research. Higher scores on the SPEAK-II indicate more knowledge about early language development.
Change in MacArthur-Bates Communication Development Inventories (MBCDI) | Baseline, 3-month follow-up, and 6-month follow-up
  The MacArthur-Bates Communication Development Inventories (MBCDI) will be given to caregivers at baseline and follow-up sessions to measure children's vocabulary. The more vocabulary words on the MBCDI that a parent reports that their child knows, the larger the child's vocabulary.

SECONDARY OUTCOMES:
Change in Self-Efficacy for Parenting Tasks-Toddler Scale | Baseline, 3-month follow-up, and 6-month follow-up
  The Self-Efficacy for Parenting Tasks-Toddler Scale will be used to assess caregivers' self-efficacy in the areas of play and teaching. The scale uses a Likert-scale to indicate how well caregivers see themselves doing a certain parenting skill. Higher scores on the Self-Efficacy Scale indicate higher levels of self-efficacy.
Change in Langauge Diversity | Baseline, 3-month follow-up, and 6-month follow-up
  To assess the quality of caregiver-child interactions, caregivers and participating children will be filmed or film themselves for a total of 10-15 minutes, at baseline, 3-month, and 6-month follow-up sessions. We will calculate the number of diverse words produced by caregivers.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatrics Department at Temple University Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alper, R.M., Luo, R., Hirsh-Pasek, K., Mogul, M., Chen, Y., Masek, L., Paterson, S., Pace, A., Adamson, L., Bakeman, R., Golinkoff, R., Owen, M. (under review). Improving child language outcomes for children in low-income households: The Duet Project.
- [Background] Baggett KM, Davis B, Feil EG, Sheeber LB, Landry SH, Carta JJ, Leve C. Technologies for expanding the reach of evidence-based interventions: Preliminary results for promoting social-emotional development in early childhood. Topics Early Child Spec Educ. 2010 Feb 1;29(4):226-238. doi: 10.1177/0271121409354782. No abstract available. PMID 20454545
- [Background] Barnard, K. E. (1998). Developing, implementing and documenting interventions with parents and young children. Zero to Three, 18(4), 23-29.
- [Background] Bedore LM, Pena ED, Summers CL, Boerger KM, Resendiz MD, Greene K, Bohman TM, Gillam RB. The measure matters: Language dominance profiles across measures in Spanish-English bilingual children. Biling (Camb Engl). 2012 Jul;15(3):616-629. doi: 10.1017/S1366728912000090. Epub 2012 Mar 20. PMID 23565049
- [Background] Birdson, D., Gertken, L.M., & Amengual, M. (2012). Bilingual Language Profile: An Easy-to-Use Instrument to Assess Bilingualism. COERLLL: University of Texas at Austin.
- [Background] Black JT, Romano PS, Sadeghi B, Auerbach AD, Ganiats TG, Greenfield S, Kaplan SH, Ong MK; BEAT-HF Research Group. A remote monitoring and telephone nurse coaching intervention to reduce readmissions among patients with heart failure: study protocol for the Better Effectiveness After Transition - Heart Failure (BEAT-HF) randomized controlled trial. Trials. 2014 Apr 13;15:124. doi: 10.1186/1745-6215-15-124. PMID 24725308
- [Background] Cartmill EA, Armstrong BF 3rd, Gleitman LR, Goldin-Meadow S, Medina TN, Trueswell JC. Quality of early parent input predicts child vocabulary 3 years later. Proc Natl Acad Sci U S A. 2013 Jul 9;110(28):11278-83. doi: 10.1073/pnas.1309518110. Epub 2013 Jun 24. PMID 23798423
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Coleman, P. K., & Karraker, K. H. (2003). Maternal self-efficacy beliefs, competence in parenting, and toddlers' behavior and developmental status. Infant Mental Health Journal, 24(2), 126-148. https://doi.org/10.1002/imhj.10048
- [Background] Dickinson, D. K., Golinkoff, R. M., & Hirsh-Pasek, K. (2010). Speaking out for language: Why language Is central to reading development. Educational Researcher, 39(4), 305-310. https://doi.org/10.3102/0013189X10370204
- [Background] Eaton WW, Muntaner C, Smith C, Tien A, Ybarra M. Center for Epidemiologic Studies Depression Scale: Review and revision (CESD and CESD-R). In: Maruish ME, ed. The Use of Psychological Testing for Treatment Planning and Outcomes Assessment. 3rd ed. Mahwah, NJ: Lawrence Erlbaum; 2004:363-377.
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Fenson, L., Pethick, S., Renda, C., Cox, J. L., Dale, P. S., & Reznick, J. S. (2000). Short-form versions of the MacArthur Communicative Development Inventories. Applied Psycholinguistics, 21(1), 95-116.
- [Background] Fernald A, Marchman VA, Weisleder A. SES differences in language processing skill and vocabulary are evident at 18 months. Dev Sci. 2013 Mar;16(2):234-248. doi: 10.1111/desc.12019. Epub 2012 Dec 8. PMID 23432833
- [Background] Goldin-Meadow S, Levine SC, Hedges LV, Huttenlocher J, Raudenbush SW, Small SL. New evidence about language and cognitive development based on a longitudinal study: hypotheses for intervention. Am Psychol. 2014 Sep;69(6):588-99. doi: 10.1037/a0036886. Epub 2014 Jun 9. PMID 24911049
- [Background] Golinkoff RM, Hoff E, Rowe ML, Tamis-LeMonda CS, Hirsh-Pasek K. Language Matters: Denying the Existence of the 30-Million-Word Gap Has Serious Consequences. Child Dev. 2019 May;90(3):985-992. doi: 10.1111/cdev.13128. Epub 2018 Aug 13. PMID 30102419
- [Background] Hammer, C.S., Scarpino, S., Cycyk, L., Sawyer, B. & Jury (2015). Center for Early Care and Education Research - Dual Language Learners (CECER-DLL) Parent Questionnaire.
- [Background] Hart, B., & Risley, T. R. (2003). The Early Catastrophe. The 30 Million Word Gap. American Educator, 27(1), 4-9.
- [Background] Hirsh-Pasek K, Adamson LB, Bakeman R, Owen MT, Golinkoff RM, Pace A, Yust PK, Suma K. The Contribution of Early Communication Quality to Low-Income Children's Language Success. Psychol Sci. 2015 Jul;26(7):1071-83. doi: 10.1177/0956797615581493. Epub 2015 Jun 5. PMID 26048887
- [Background] Hoff, E. (2006). How social contexts support and shape language development. Developmental Review, 26(1), 55-88. https://doi.org/10.1016/j.dr.2005.11.002
- [Background] Hoff E. Interpreting the early language trajectories of children from low-SES and language minority homes: implications for closing achievement gaps. Dev Psychol. 2013 Jan;49(1):4-14. doi: 10.1037/a0027238. Epub 2012 Feb 13. PMID 22329382
- [Background] Knauer, H. A., Ozer, E. J., Dow, W. H., & Fernald, L. C. H. (2018). Parenting quality at two developmental periods in early childhood and their association with child development. Early Childhood Research Quarterly. https://doi.org/10.1016/j.ecresq.2018.08.009
- [Background] Luo R, Alper RM, Hirsh-Pasek K, Mogul M, Chen Y, Masek LR, Paterson S, Pace A, Adamson LB, Bakeman R, Golinkoff RM, Owen MT. Community-Based, Caregiver-Implemented Early Language Intervention in High-Risk Families: Lessons Learned. Prog Community Health Partnersh. 2019;13(3):283-291. doi: 10.1353/cpr.2019.0056. PMID 31564669
- [Background] Luo, R., & Tamis-LeMonda, C. S. (2017). Reciprocity between maternal questions and child contributions during book-sharing. Early Childhood Research Quarterly, 38, 71-83. https://doi.org/10.1016/j.ecresq.2016.08.003
- [Background] MacWhinney, B. (2000). The CHILDES Project: Tools for analyzing talk. (3rd Edition). Mahwah, NJ: Lawrence Erlbaum Associates.
- [Background] Miller, J. & Iglesias, A. (2017). Systematic Analysis of Language Transcripts (SALT), Research Version 18 [Computer Software]. Madison, WI: SALT Software, LLC.
- [Background] Murphey, D., Epstein, D., Shaw, S., McDaniel, T., & Steber, K. (2018). The status of infants and toddlers in Philadelphia. Child Trends. Retrieved from https://www.childtrends.org/wp-content/uploads/2018/08/PhiladelphiaInfantandToddlers_ChildTrends_September2018.pdf
- [Background] Pace, A., Alper, R., Burchinal, M. R., Golinkoff, R. M., & Hirsh-Pasek, K. (2018). Measuring success: Within and cross-domain predictors of academic and social trajectories in elementary school. Early Childhood Research Quarterly. https://doi.org/10.1016/j.ecresq.2018.04.001
- [Background] Peña, Guitierrez-Clellan, Igelsias, Goldstein, & Bedore (2018). Bilingual English-Spanish Assessment (BESA). Brookes Publishing.
- [Background] Pew Charitable Trusts. (2017). Philadelphia's poor: Who they are, where they live, and how that's changed. Retrieved from https://www.pewtrusts.org/- /media/assets/2017/11/pri_philadelphias_poor.pdf
- [Background] Powell, D. R., Diamond, K. E., Burchinal, M. R., & Koehler, M. J. (2010). Effects of an early literacy professional development intervention on head start teachers and children. Journal of Educational Psychology, 102(2), 299-312. https://doi.org/10.1037/a0017763
- [Background] Radloff, L. (1977). The CES-D Scale: A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement, 1(3), 385-401.
- [Background] Romeo RR, Leonard JA, Robinson ST, West MR, Mackey AP, Rowe ML, Gabrieli JDE. Beyond the 30-Million-Word Gap: Children's Conversational Exposure Is Associated With Language-Related Brain Function. Psychol Sci. 2018 May;29(5):700-710. doi: 10.1177/0956797617742725. Epub 2018 Feb 14. PMID 29442613
- [Background] Rowe ML. A longitudinal investigation of the role of quantity and quality of child-directed speech in vocabulary development. Child Dev. 2012 Sep-Oct;83(5):1762-74. doi: 10.1111/j.1467-8624.2012.01805.x. Epub 2012 Jun 20. PMID 22716950
- [Background] Rowe ML, Leech KA, Cabrera N. Going Beyond Input Quantity: Wh-Questions Matter for Toddlers' Language and Cognitive Development. Cogn Sci. 2017 Feb;41 Suppl 1:162-179. doi: 10.1111/cogs.12349. Epub 2016 Feb 29. PMID 26923546
- [Background] Song L, Spier ET, Tamis-Lemonda CS. Reciprocal influences between maternal language and children's language and cognitive development in low-income families. J Child Lang. 2014 Mar;41(2):305-26. doi: 10.1017/S0305000912000700. Epub 2013 Jan 30. PMID 23360640
- [Background] Sperry DE, Sperry LL, Miller PJ. Reexamining the Verbal Environments of Children From Different Socioeconomic Backgrounds. Child Dev. 2019 Jul;90(4):1303-1318. doi: 10.1111/cdev.13072. Epub 2018 Apr 30. PMID 29707767
- [Background] Spring B, Schneider K, McFadden HG, Vaughn J, Kozak AT, Smith M, Moller AC, Epstein LH, Demott A, Hedeker D, Siddique J, Lloyd-Jones DM. Multiple behavior changes in diet and activity: a randomized controlled trial using mobile technology. Arch Intern Med. 2012 May 28;172(10):789-96. doi: 10.1001/archinternmed.2012.1044. PMID 22636824
- [Background] Squires, J., Bricker, D., Twombly, E., Nickel, R., Clifford, J., Murphy, K., … Farrell, J. (2009). Ages and Stages Questionnaire-Third Edition. Brookes Publishing Co.
- [Background] Suskind DL, Leung CYY, Webber RJ, Hundertmark AC, Leffel KR, Fuenmayor Rivas IE, Grobman WA. Educating Parents About Infant Language Development: A Randomized Controlled Trial. Clin Pediatr (Phila). 2018 Jul;57(8):945-953. doi: 10.1177/0009922817737079. Epub 2017 Oct 26. PMID 29073768
- [Background] Tamis-LeMonda, C. S., Kuchirko, Y., & Song, L. (2014). Why is infant language learning facilitated by parental responsiveness? Current Directions in Psychological Science, 23(2), 121-126. https://doi.org/10.1177/0963721414522813
- [Background] Uccelli P, Demir-Lira OE, Rowe ML, Levine S, Goldin-Meadow S. Children's Early Decontextualized Talk Predicts Academic Language Proficiency in Midadolescence. Child Dev. 2019 Sep;90(5):1650-1663. doi: 10.1111/cdev.13034. Epub 2018 Jan 23. PMID 29359315
- [Background] Varney JE, Weiland TJ, Inder WJ, Jelinek GA. Effect of hospital-based telephone coaching on glycaemic control and adherence to management guidelines in type 2 diabetes, a randomised controlled trial. Intern Med J. 2014 Sep;44(9):890-7. doi: 10.1111/imj.12515. PMID 24963611
- [Background] Vismara LA, McCormick C, Young GS, Nadhan A, Monlux K. Preliminary findings of a telehealth approach to parent training in autism. J Autism Dev Disord. 2013 Dec;43(12):2953-69. doi: 10.1007/s10803-013-1841-8. PMID 23677382
- [Background] Wainer AL, Ingersoll BR. Increasing Access to an ASD Imitation Intervention Via a Telehealth Parent Training Program. J Autism Dev Disord. 2015 Dec;45(12):3877-90. doi: 10.1007/s10803-014-2186-7. PMID 25035089
- [Background] Zimmerman, I. L., Steiner, V. G., & Pond, R. E. (2012). Preschool Language Scales, Fifth Edition Screening Test English and Spanish (PLS-5). Pearson Clinical.